CLINICAL TRIAL: NCT02220985
Title: A Phase II Study Evaluating Selective Depletion of CD45RA+ T Cells From Allogeneic Peripheral Blood Stem Cell Grafts From HLA-Matched Related and Unrelated Donors for Prevention of GVHD
Brief Title: Selective Depletion of CD45RA+ T Cells From Allogeneic Peripheral Blood Stem Cell Grafts From HLA-Matched Related and Unrelated Donors in Preventing GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2684.00; NCI-2014-01301 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2684.00 (Other: Fred Hutch/University of Washington Cancer Consortium); R01HL121568 (NIH); RG9214012 (Other: Fred Hutch/University of Washington Cancer Consortium); 2P01CA018029 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Biphenotypic Leukemia; Acute Leukemia of Ambiguous Lineage; Acute Undifferentiated Leukemia; Allogeneic Hematopoietic Stem Cell Transplant Recipient; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blastic Plasmacytoid Dendritic Cell Neoplasm; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Donor; Lymphoblastic Lymphoma; Myelodysplastic Syndrome With Excess Blasts; Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome With Excess Blasts-2; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Blast Crisis; Blastic Plasmacytoid Dendritic Cell Neoplasm; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cyclophosphamide; fludarabine phosphate; Methotrexate; merphos; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (MRD) (Experimental): HIGH-INTENSITY MYELOABLATIVE CONDITIONING: Patients undergo total body irradiation BID on days -10 to -7. Patients also receive thiotepa IV over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  TRANSPLANT: In all arms, patients undergo allogeneic HSCT with GCSF-mobilized CD34-enriched PBSC and CD45RA-depleted cells on day 0.
  GVHD PROPHYLAXIS: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or PO (BID if given PO) for 50 days with taper in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation
- Arm B (MRD) (Experimental): LOWER-INTENSITY MYELOABLATIVE CONDITIONING: Patients receive cyclophosphamide IV over 1 hour on day -6, fludarabine phosphate IV over 30 minutes on days -6 to -2, and thiotepa IV over 4 hours on days -5 and -4. Patients also undergo total body irradiation QD on days -2 and -1.
  TRANSPLANT: In all arms, patients undergo allogeneic HSCT with GCSF-mobilized CD34-enriched PBSC and CD45RA-depleted cells on day 0.
  GVHD PROPHYLAXIS: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or PO (BID if given PO) for 50 days and mycophenolate mofetil IV and PO every 8 hours on day -3 to approximately day 30, with or without taper at the discretion of the treating physician. Mycophenolate mofetil should be continued or resumed after day 30 if donor chimerism is low, after discussion with the Principal Investigator.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation
- Arm C (MUD) (Experimental): HIGH-INTENSITY MYELOABLATIVE CONDITIONING: Patients undergo total body irradiation BID on days -10 to -7. Patients also receive thiotepa IV over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  TRANSPLANT: In all arms, patients undergo allogeneic HSCT with G-CSF-mobilized CD34-enriched PBSC and CD45RA-depleted cells on day 0.
  GVHD PROPHYLAXIS: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or PO (BID if given PO) for 50 days with taper in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation
- Arm D (MUD) (Experimental): LOWER-INTENSITY MYELOABLATIVE CONDITIONING: Patients receive cyclophosphamide IV over 1 hour on day -6, fludarabine phosphate IV over 30 minutes on days -6 to -2, and thiotepa IV over 4 hours on days -5 and -4. Patients also undergo total body irradiation QD on days -2 and -1.
  TRANSPLANT: In all arms, patients undergo allogeneic HSCT with G-CSF-mobilized CD34-enriched PBSC and CD45RA-depleted cells on day 0.
  GVHD PROPHYLAXIS: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or PO (BID if given PO) for 50 days and mycophenolate mofetil IV and PO every 8 hours on day -3 to approximately day 30, with or without taper at the discretion of the treating physician. Mycophenolate mofetil should be continued or resumed after day 30 if donor chimerism is low, after discussion with the Principal Investigator.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Thiotepa

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm A (MRD); Arm C (MUD)
Drug: Mycophenolate Mofetil — Given IV and PO
  Other Names: Cellcept; MMF
  Arms: Arm B (MRD); Arm D (MUD)
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSCT with GCSF-mobilized CD34-enriched PBSC
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSCT with CD45RA-depleted cells
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation; TBI; Whole Body Irradiation
  Arms: Arm A (MRD); Arm B (MRD); Arm C (MUD)

SUMMARY:
This phase II trial is for patients with acute lymphocytic leukemia, acute myeloid leukemia, myelodysplastic syndrome or chronic myeloid leukemia who have been referred for a peripheral blood stem cell transplantation to treat their cancer. In these transplants, chemotherapy and total-body radiotherapy ('conditioning') are used to kill residual leukemia cells and the patient's normal blood cells, especially immune cells that could reject the donor cells. Following the chemo/radiotherapy, blood stem cells from the donor are infused. These stem cells will grow and eventually replace the patient's original blood system, including red cells that carry oxygen to our tissues, platelets that stop bleeding from damaged vessels, and multiple types of immune-system white blood cells that fight infections. Mature donor immune cells, especially a type of immune cell called T lymphocytes (or T cells) are transferred along with these blood-forming stem cells. T cells are a major part of the curative power of transplantation because they can attack leukemia cells that have survived the chemo/radiation therapy and also help to fight infections after transplantation. However, donor T cells can also attack a patient's healthy tissues in an often-dangerous condition known as Graft-Versus-Host-Disease (GVHD). Drugs that suppress immune cells are used to decrease the severity of GVHD; however, they are incompletely effective and prolonged immunosuppression used to prevent and treat GVHD significantly increases the risk of serious infections. Removing all donor T cells from the transplant graft can prevent GVHD, but doing so also profoundly delays infection-fighting immune reconstitution and eliminates the possibility that donor immune cells will kill residual leukemia cells. Work in animal models found that depleting a type of T cell, called naïve T cells or T cells that have never responded to an infection, can diminish GVHD while at least in part preserving some of the benefits of donor T cells including resistance to infection and the ability to kill leukemia cells. This clinical trial studies how well the selective removal of naïve T cells works in preventing GVHD after peripheral blood stem cell transplants. This study will include patients conditioned with high or medium intensity chemo/radiotherapy who can receive donor grafts from related or unrelated donors.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 4 treatment arms.

CONDITIONING:

ARMS A AND C (high-intensity myeloablative conditioning): Patients undergo total body irradiation twice daily (BID) on days -10 to -7. Patients also receive thiotepa intravenously (IV) over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.

ARMS B AND D (lower-intensity myeloablative conditioning): Patients receive cyclophosphamide IV over 1 hour on day -6, fludarabine phosphate IV over 30 minutes on days -6 to -2, and thiotepa IV over 4 hours on days -5 and -4. Patients also undergo total body irradiation once daily (QD) on days -2 and -1.

TRANSPLANT: In all arms, patients undergo allogeneic HSCT with granulocyte colony-stimulating factor (GCSF)-mobilized CD34-enriched PBSC and CD45RA-depleted cells on day 0.

GVHD PROPHYLAXIS:

ARMS A AND C: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or orally (PO) (BID if given PO) for 50 days with taper in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

ARMS B AND D: Beginning day -1, patients receive tacrolimus IV over 22-24 hours or PO (BID if given PO) for 50 days and mycophenolate mofetil IV and PO every 8 hours on days -3 to approximately day 30, with or without taper at the discretion of the treating physician. Mycophenolate mofetil should be continued or resumed after day 30 if donor chimerism is low, after discussion with the principal investigator.

After completion of study treatment, patients are followed up at 80-100 days, 360 days, and then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered appropriate candidates for allogeneic hematopoietic stem cell transplantation and have one of the following diagnoses:

  * Acute lymphocytic leukemia in first or subsequent remission
  * Acute myeloid leukemia in first or subsequent remission
  * Acute lymphocytic leukemia in relapse or primary refractory disease with a circulating blast count of no more than 10,000/mm^3 (Arms A or C only)
  * Acute myeloid leukemia in relapse or primary refractory disease with a circulating blast count of no more than 10,000/mm^3 (Arms A or C only)
  * Refractory anemia with excess blasts (RAEB-1 and RAEB-2) (if the patient has received previous induction chemotherapy within 60 days)
  * Chronic myelogenous leukemia with a history of accelerated phase or blast crisis (if the patient has received at least one course of induction chemotherapy)
  * Other acute leukemia or related neoplasm (including but not limited to 'biphenotypic', 'undifferentiated' or 'ambiguous lineage' acute leukemia, blastic plasmacytoid dendritic cell neoplasm or lymphoblastic lymphoma)
* Patients 0-49 years old will be enrolled in Arm A or C (high-intensity)
* Patients 50-60 years old will be enrolled in Arm B or D (lower intensity); patients eligible for Arms B or D also include those who have received previous allogeneic HCT, or who have co-morbid conditions rendering them unsuitable for high-dose conditioning, determined in consultation with the principal investigator
* Patient with a HLA-matched (HLA-A, B, C, and DR beta 1 [DRB1] molecularly matched) unrelated donor or related donor capable of donating PBSC
* DONOR INCLUSION:
* HLA-matched related donors >= 18 years and capable and willing to donate PBSC (Arms A and B)
* HLA-matched unrelated donors (HLA-A, B, C, and DRB1 matched based on high-resolution typing) capable and willing to donate PBSC (Arms C and D)

Exclusion Criteria:

* Patients with central nervous system (CNS) involvement refractory to intrathecal chemotherapy and/or standard cranial-spinal radiation
* Patients on other experimental protocols for prevention of acute GVHD
* Patient weight >= 100 kg; patients >= 70 kg with MUDs must be discussed with the principal investigator
* Patients who are human immunodeficiency virus positive (HIV+)
* Patients with uncontrolled infections for whom myeloablative HCT is considered contraindicated by the consulting infectious disease physician (upper respiratory tract viral infection does not constitute an uncontrolled infection in this context)
* Patients with organ dysfunction
* ARM A OR C EXCLUSION:
* Creatinine > 1.5 mg/dl at the present time; patients with a known history of creatinine > 1.5 mg/dl must have a current estimated creatinine clearance of > 40 ml/min
* Cardiac ejection fraction < 45%
* Diffusing capacity of the lung for carbon monoxide (DLCO) corrected < 60%; patients who are unable to perform pulmonary function tests (for example, due to young age and/or developmental status) will be excluded if the oxygen (O2) saturation is < 92% on room air
* Liver function abnormality; patients who have liver function tests (LFTs) (including total bilirubin, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) >= twice the upper limit of normal should be evaluated by a gastrointestinal (GI) physician; unless there is a clear precipitating factor (such as an azole, methotrexate, Bactrim or another drug); if the GI physician considers that HCT on the high-intensity arms of protocol is contraindicated for that patient the patient may be considered for treatment on the lower intensity arm of the protocol or excluded from the protocol; patients with Gilbert's syndrome and no other known liver function abnormality and patients with reversible drug-related transaminitis do not necessarily require GI consultation and may be included on the high-intensity arms of the protocol
* ARM B OR D EXCLUSION:
* Creatinine > 2.0 mg/dl at the present time; patients with a known history of creatinine > 1.5 mg/dl must have a current estimated creatinine clearance > 40 ml/min
* Cardiac ejection fraction < 35%
* DLCO corrected < 50%; patients who are unable to perform pulmonary function tests (for example, due to young age and/or developmental status) will be excluded if the O2 saturation is < 92% on room air; patients with a DLCO 50-60% must also have a partial pressure of oxygen (pO2) of > 80 mmHg
* Liver function abnormality; patients who have LFTs >= twice the upper limit of normal should be evaluated by a GI physician unless there is a clear precipitating factor (such as an azole, methotrexate, Bactrim or another drug); patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Patients will be excluded from Arms A and C if they have received a previous myeloablative transplant; patients who have received a prior HCT at least 6 months prior may be considered for inclusion on Arms B or D after discussion with the principal investigator (PI)
* Patients with a life expectancy < 3 months from co-existing disease other than the leukemia or RAEB
* Patients who are pregnant or breast-feeding
* Fertile patients of child bearing age unwilling to use contraception during and for 12 months post-transplant
* Patients with a significant other medical conditions that would make them unsuitable for transplant
* Patients with a known hypersensitivity to tacrolimus, methotrexate (Arm A or C) or MMF (Arm B or D)
* DONOR EXCLUSION:
* Donors who are HIV-1, HIV-2, human T-lymphotropic virus (HTLV)-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection
* Donors who fail eligibility requirements for donation of cells or tissue for donation of a Human Cell and Tissue Products (HCT/P) will be excluded unless use of the cells complies urgent medical need or allogeneic use in a first-degree or second-degree relative
* Unrelated donors donating outside of the United States of America (USA)

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of chronic graft-versus-host disease (GHVD), defined operationally as the occurrence of compatible symptoms meeting National Institutes of Health criteria and requiring systemic pharmacological immunosuppression | Up to 5 years
  Match related donor (MRD)-high intensity (Arm A), MRD-lower intensity (Arm B), match unrelated donor (MUD)-high intensity (Arm C) and MUD-lower intensity (Arm D) cohorts will be analyzed separately.
Use of additional immune suppressive agents other than first line therapy (prednisone and tacrolimus/cyclosporine) | Up to 5 years
Time to completion of prednisone | Up to 5 years
Time to completion of all immunosuppression | Up to 5 years
Requirement of immunosuppression after transplant | At 2 years after transplant
Presence of acute graft-versus-host disease (GVHD) grades II-IV | Up to day 100
  Defined operationally as the occurrence of compatible symptoms or signs in the skin, gastrointestinal tract, or liver.
Requirement for secondary systemic therapy for acute graft-versus-host disease (GVHD) management | Up to day 100
Graft failure | Up to day 28
  Defined operationally as failure to reach an absolute neutrophil count (ANC) of > 500/ul for 3 consecutive days by day 28 or irreversible decrease in ANC to < 100 after an established donor graft.

SECONDARY OUTCOMES:
Time to absolute neutrophil count (ANC) of > 500/uL on the first of three consecutive days | Up to 5 years
Time to absolute neutrophil count (ANC) of > 1,000/uL on the first of three consecutive test results | Up to 5 years
Time to platelet count > 20,000/uL for 3 days without transfusion | Up to 5 years
Time to platelet count > 50,000/uL for 3 days without transfusion | Up to 5 years
Chimerism analysis | Up to 360 days
  Will be analyzed from peripheral blood or marrow.
Relapse | Up to 5 years
  Defined by the presence of malignant cells in marrow, peripheral blood, or extramedullary sites by histopathology.
Transplant related mortality | Up to 5 years
  Defined as mortality in any patient for whom there has not been a diagnosis of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bleakley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Bleakley M, Sehgal A, Seropian S, Biernacki MA, Krakow EF, Dahlberg A, Persinger H, Hilzinger B, Martin PJ, Carpenter PA, Flowers ME, Voutsinas J, Gooley TA, Loeb K, Wood BL, Heimfeld S, Riddell SR, Shlomchik WD. Naive T-Cell Depletion to Prevent Chronic Graft-Versus-Host Disease. J Clin Oncol. 2022 Apr 10;40(11):1174-1185. doi: 10.1200/JCO.21.01755. Epub 2022 Jan 10. PMID 35007144